CLINICAL TRIAL: NCT02580422
Title: Pilot Project for Cardiopulmonary and Functional Evaluation in Patients With Pancreatic Cancer Associated Cachexia
Status: Terminated | Type: Observational
Why Stopped: Low accrual
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Safi Shahda, Assistant Professor of Clinical Medicine, Indiana University
Other Study IDs: IUSCC-0547
Record Dates: First submitted 2015-10-06; First posted 2015-10-20 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Cachexia; Pancreatic Cancer
Keywords: Echocardiography
MeSH Terms: conditions — Cachexia; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected: one sample for cytokine analysis, one sample for future research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cachexia is a systemic catabolic syndrome with apparent effect on skeletal muscles, tolerance to chemotherapy, early toxicity and quality of life; however, its effect on cardiopulmonary function is not well understood. Preclinical studies demonstrated diaphragmatic muscle wasting(29) and left ventricular wasting and fibrosis associated with mouse cachexia models.(40) Many patients, who experience cancer cachexia, describe a generalized debility and a sense of breathlessness(41) despite adequate oxygenation in the peripheral blood as measured by pulse oximetry. Whether this is related to deconditioning associated with chemotherapy or related to direct effect on cardiac and diaphragmatic muscles remains unknown. In this pilot study, the investigators propose to perform a preliminary evaluation of the cardiopulmonary function in patients with pancreatic cancer, who are likely to develop cachexia, to assess for the feasibility of performing a larger prospective study to understand the impact of cancer cachexia on cardiopulmonary function. This pilot study will provide the foundation to potentially identify cachexia in early stages (pre-cachexia) to develop pharmacological or exercise based interventions to prevent or delay its progression. Based on clinical experience and published literature, it is expected that 60-70% of patients will have >10% weight loss during the course of this disease. More commonly, this is associated with clinical or radiographic disease progression, but certainly it can happen throughout the course of the disease even without disease progression.

DETAILED DESCRIPTION:
Primary Objective:

To assess the feasibility of performing a prospective cardiopulmonary and physical function assessment in patients with advanced pancreatic ductal adenocarcinoma (PDAC) who are expected to develop cachexia.

Secondary Objectives:

1. To measure the changes in maximal expiratory pressure (MEP) and maximal inspiratory pressure (MIP) in patients with progressive PDAC and/or cancer associated cachexia
2. To measure changes in strain echocardiography in patients with progressive PDAC and/or cancer associated cachexia
3. To assess functional changes in patients with progressive PDAC and/or cancer associated cachexia
4. To assess body composition changes associated with cachexia or disease progression
5. To measure the levels of cytokines from peripheral blood in patients with cachexia

Procedures:

All study procedures will be done at two time points (T1=baseline or study entry, T2=at disease progression or development of cachexia). Patients will undergo echocardiography with strain evaluation at Indiana University Health Echocardiography Laboratory and pulmonary function tests as per institutional guidelines at IUH PFT laboratory at University Hospital. Patients will also have 20mL (2 red top tubes) of blood drawn for the studies outlined in Section 7.5. Standard of care labs will be taken from the patient's medical records. Patients also will be evaluated using three standardized functional assessment tools commonly utilized in physical rehabilitation: 1) 5 Times Sit-to-Stand Test; 2) 6 Minute Walk Test; and 3) grip dynamometry. Standard of care CT scan obtained at the time of tumor assessment will enable the investigators to assess body muscle mass as described in Section 7.4. In addition, the investigators will administer three standardized survey tools to assess quality of life and prior level of function: 1) The Short Form 36 (SF-36); 2) Lower Extremity Functional Scale (LEFS); and 3) Scored Patient-Generated Subjective Global Assessment (PG-SGA).

Sample Size:

Due to the risk of clinical deterioration or drop out of the study and inability to undergo T2 evaluation, the investigators will plan on enrolling 133% of desired number of subjects, accounting for 33% missing T2 data. This is likely a high number; however, this will enable data collection from 12-15 patients at both time points and all proposed tests.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with locally advanced, metastatic or recurrent pancreatic ductal adenocarcinoma (PDAC)
2. Patients who are being treated and/or followed at Indiana University Simon Cancer Center or Eskenazi Hospital
3. ECOG PS 0-2 at the time of study enrollment
4. Life expectancy > 6 months
5. Adequate organ function

   * As defined by the following laboratory values at study entry:
   * Hemoglobin ≥ 9 g/dL (transfusions are acceptable)
   * ANC ≥ 1.5 x 109/L
   * Platelets ≥ 100 x 109/L
   * Creatinine ≤ 1.5 x ULN, or creatinine clearance ≥ 50 mL/min (estimated by Cockcroft-Gault or measured)
   * Total bilirubin ≤ 1.5 x ULN
   * AST/ALT ≤ 3 x ULN
6. Willingness to sign informed consent and to perform pulmonary function tests (PFTs) and strain echocardiogram

Exclusion Criteria:

1. Known history of congestive heart failure (NYHA class III or IV)
2. Reported weight loss more than 10% within 3 months prior to study entry
3. Known history of pulmonary disease such as pulmonary hypertension, chronic obstructive pulmonary disease requiring medical management or previous lung resection
4. Current liver cirrhosis
5. Current chronic kidney disease
6. Inability or refusal to receive systemic therapy
7. Inability to comply with pulmonary function tests (PFTs)
8. Large volume ascites interfering with ability of respiration
9. Current unstable angina (or history of within last 6 months)
10. Recent myocardial infraction (within last 6 months)
11. Recent pneumothorax (within last 6 months)
12. Uncontrolled hypertension (per investigator's discretion)
13. Lung biopsy within one week from PFT
14. Recent surgery < 4 weeks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential participants will be identified from the outpatient oncology clinic at the Indiana University Health Melvin and Bren Simon Cancer Center or Sidney & Lois Eskenazi Health Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-05-27 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
The number of patients who have changes in echocardiography, pulmonary function or one or more part of their functional evaluation tests | Baseline to disease progression or development of cachexia (approximately 6 months)
  Changes are significant if they are > 15% from baseline. Development of cachexia is defined by ≥ 10% of weight loss from baseline.

SECONDARY OUTCOMES:
Change in pulmonary function | Baseline to disease progression or development of cachexia (approximately 6 months)
  Measured by comparing scores (maximal expiratory pressure [MEP] and maximal inspiratory pressure [MIP]) from forced spirometry with folow volume loop test.
Change in strain echocardiogram | Baseline to disease progression or development of cachexia (approximately 6 months)
  Measured by comparing strain echocardiograms
Change in self-reported quality of life | Baseline to disease progression or development of cachexia (approximately 6 months)
  Measured by comparing Short Form-36 questionnaire scores
Change in self-reported function via LEFS questionnaire | Baseline to disease progression or development of cachexia (approximately 6 months)
  Measured by comparing Lower Extremity Functional Scale (LEFS) questionnaire scores
Change in self-reported function via PG-SGA questionnaire | Baseline to disease progression or development of cachexia (approximately 6 months)
  Measured by comparing Patient-Generated Subjective Global Assessment (PG-SGA) questionnaire scores
Change in functional evaluation test | Baseline to disease progression or development of cachexia (approximately 6 months)
  Measured by comparing grip dynamometry, 6-minute walk test, 5-minute sit-to-stand test scores
Change in body composition via CT scan | Baseline to disease progression or development of cachexia (approximately 6 months)
  Measured by comparing CT scans that are analyzed using Sliceomatic (Tomovision) technology
Change in levels of cytokines | Baseline to disease progression or development of cachexia (approximately 6 months)
  Measured through blood samples collected at each time point which are evaluated for cytokine levels using enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Safi Shahda, MD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (2):
- United States (2):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney & Lois Eskenazi Hospital, Indianapolis, Indiana

REFERENCES:
- [Background] Roberts BM, Ahn B, Smuder AJ, Al-Rajhi M, Gill LC, Beharry AW, Powers SK, Fuller DD, Ferreira LF, Judge AR. Diaphragm and ventilatory dysfunction during cancer cachexia. FASEB J. 2013 Jul;27(7):2600-10. doi: 10.1096/fj.12-222844. Epub 2013 Mar 20. PMID 23515443
- [Background] Muhlfeld C, Das SK, Heinzel FR, Schmidt A, Post H, Schauer S, Papadakis T, Kummer W, Hoefler G. Cancer induces cardiomyocyte remodeling and hypoinnervation in the left ventricle of the mouse heart. PLoS One. 2011;6(5):e20424. doi: 10.1371/journal.pone.0020424. Epub 2011 May 26. PMID 21637823
- [Background] Coats AJ. Origin of symptoms in patients with cachexia with special reference to weakness and shortness of breath. Int J Cardiol. 2002 Sep;85(1):133-9. doi: 10.1016/s0167-5273(02)00242-5. PMID 12163218